CLINICAL TRIAL: NCT06510998
Title: Effectiveness and Mechanisms of Isometric Resistance Exercise to Reduce Blood Pressure in a Chinese Population: a Randomized-controlled Trial
Brief Title: Isometric Resistance Exercise for Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, clinical associate professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022.618
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric exercise (Experimental): 2 minutes wall squat, with 2 minutes rest between sets
  * to perform 4 sets in total/day
  * at least 3 days/week
  * totally for 24-weeks
  Interventions: Behavioral: isometric wall exercise
- passive stretching (Active Comparator): 14 minutes passive stretching
  * at least 3 days/week
  * totally 24-weeks
  Interventions: Behavioral: passive stretching

INTERVENTIONS:
Behavioral: isometric wall exercise — Each exercise session will contain 4 sets of 2-minute wall squat isometric holds with 2 minutes of rest between each set (approximately 14 minutes per session in total), and a total of 3 sessions will be arranged every week (with ideally 48 h between exercises)
  Arms: Isometric exercise
Behavioral: passive stretching — A frequency-matched (3x/week) and time-matched (~14 minutes each session) passive static stretching exercise will be used
  Arms: passive stretching

SUMMARY:
Background: Isometric resistance exercises (IREs) have great potential to improve blood pressure (BP) control. However, the effectiveness of IREs in reducing HT is still unknown because their hypotensive effects have not been detected using ambulatory BP measurements (ABPM), which are the current standard for BP measurement.

Methods: This first adequately-powered RCT will involve 390 patients with HT who do not meet the current physical activity guidelines defined by the World Health Organization. Participants will be randomly assigned in a 1:1 ratio using stratified and blocked randomization to either the IRE (wall squat) group or stretching exercise (active control) group. A well-structured, widely accepted, and validated 24-week wall squat program (2 minutes per exercise, 2 minutes of rest between sets, and 3 sessions per week) will be implemented, as it has been commonly used in previous research. Adherence to the program will be monitored using smartwatches, and regular contact with patients through social media will help ensure adherence. All patients will be followed up for 1 year to investigate the long-term effects of IREs on BP. Control group will receive exact same treatment except that IRE is replaced by frequency-matched and time-matched stretching exercise. The primary outcome measure will be systolic daytime ABPM BP at 24 weeks. Secondary outcome measures will include other BP and ABPM parameters at 12 weeks, 24weeks and 1year, cfPWV at baseline, 24 weeks and 1year, and FMD at baseline and 24weeks. Safety data will be collected and reported.

ELIGIBILITY:
Inclusion Criteria:

* a suboptimal daytime SBP of >135-160 mmHg on a 24-h ABPM
* reported no regular physical activity or less than that recommended for adults by the World Health Organization (e.g. <150 minutes of moderate-intensity aerobic exercise per week)
* on stable doses of anti-HT medication(s) for ≥4 weeks if the patient is receiving drug treatments;
* agree for no drug changes during the intervention period (24 weeks);

Exclusion Criteria:

* cannot provide informed consent
* unwillingness to repeat ABPM
* relative contraindications to ABPM (i.e. diagnosed atrial fibrillation, nighttime workers, occupational drivers, or patients with bleeding tendencies)
* severe osteoarthritis pending knee replacement surgery
* known secondary HT
* use of ≥3 anti-HT medications at maximum doses or ≥4 anti-HT medications
* SBP or DBP are >160 mmHg or >100 mmHg, respectively, on ABPM at baseline or at 12 weeks follow-up to ensure safety
* pregnancy/breastfeeding
* active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-07-28 (Estimated); Study Completion 2027-09-28 (Estimated)

PRIMARY OUTCOMES:
daytime systolic blood pressure (BP) assessed via ambulatory blood pressure monitoring (ABPM) | 24-week after recruitment (immediate post-intervention)
  systolic blood pressure (SBP) measured from a 24-h ABPM

SECONDARY OUTCOMES:
Other blood pressure indices | 24-week, 1 year
  other BP indices from ABPM (i.e. daytime diastolic BP [DBP] at 24-week, daytime SBP/DBP at 1 year, and 24-hour and nighttime SBP and DBP at 24-week and 1 year)
Carotid-femoral pulse wave velocity | 24-week after recruitment (immediate post-intervention), 1 year
  This will be analysed by applanation tonometry using SphygmoCor (AtCor Medical Pty Ltd) with the accompanying SphygmoCor Software Suite (SphygmoCor System
flow-mediated dilation of brachial artery (FMD) | 24-week after recruitment (immediate post-intervention), 1 year
  The longitudinal image of brachial artery is obtained 5-10cm above the elbow using a high frequency linear array vascular transducer XL14 (Philips Medical Systems, Bothell, WA, USA). After a qualified image is acquired for analysis, a pressure cuff placed distal to the imaging probe at the forearm will be inflated to 50mmHg above the systolic pressure for 5 minutes. The longitudinal image of the brachial artery is scan continuous for 3 minutes after the deflation of the cuff. Due to budget limitations, only the first 100 (50 intervention and 50 control) patients with receive FMD

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Lek Yuen General Outpatient Clinic, Hong Kong
  - School of public health and primary care, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes